CLINICAL TRIAL: NCT05885464
Title: A Phase 1/2, Dose-Exploration and Dose-Expansion Study Evaluating the Safety and Efficacy of Multiplex Base-Edited, Allogeneic Anti-CD7 CAR-T Cells (BEAM-201) in Relapsed/Refractory T-Cell Acute Lymphoblastic Leukemia (T-ALL) or T-Cell Lymphoblastic Lymphoma (T-LL)
Brief Title: A Study Evaluating the Safety and Efficacy of BEAM-201 in Relapsed/Refractory T-Cell Acute Lymphoblastic Leukemia (T-ALL) or T-Cell Lymphoblastic Lymphoma (T-LL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beam Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTX-ALO-001
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Lymphoblastic Lymphoma; T-Cell Lymphoblastic Leukemia/Lymphoma; Lymphoblastic Leukemia
Keywords: Lymphoblastic Leukemia; Lymphoblastic Lymphoma; Base editing; CAR-T
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma

STUDY DESIGN:
Intervention Model Description: The maximum number of patients for this study is approximately 102 patients:
  * 36 patients in the Phase 1 dose exploration
  * approximately 12 patients in the Phase 1 dose-expansion cohorts
  * 6 patients in the pediatric cohort
  * approximately 48 patients in the Phase 2 cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fludarabine, cyclophosphamide and alemtuzumab (Experimental): Lymphodepletion regimen including fludarabine, cyclophosphamide and alemtuzumab
  Interventions: Biological: BEAM-201
- Fludarabine, cyclophosphamide without alemtuzumab (Experimental): Lymphodepletion regimen without Alz but consisting of the same dose of Flu/Cy as in the other arm
  Interventions: Biological: BEAM-201

INTERVENTIONS:
Biological: BEAM-201 — A single dose of BEAM-201 administered by IV following one of two lymphodepletion regimens

SUMMARY:
This is a Phase 1/2, multicenter, open-label study to evaluate the safety and efficacy of BEAM-201 in patients with relapsed/refractory T-ALL or T-LL. This study consists of Phase 1 dose-exploration cohorts, Phase 1 dose-expansion cohort(s), a Phase 1 pediatric cohort (will enroll patients ages 1 to < 12 years), and a Phase 2 cohort.

ELIGIBILITY:
Key Inclusion Criteria:

1. Ages 18 to ≤ 50 years.
2. Ages ≥ 1 year to < 18 years, after health authority approval.
3. T-ALL/T-LL that is CD7-positive (defined as at least 20% of blasts positive for CD7 by flow cytometry or immunohistochemistry based on assessment of the study site's CLIA [Clinical Laboratory Improvement Amendments of 1988] certified facility) in second or greater relapse, first relapse post-transplant relapse, or chemotherapy-refractory disease. Specifically:

   1. Second or greater relapse or post-transplant relapse, defined as:

      * BM with ≥ 5% lymphoblasts by morphologic assessment or evidence of extramedullary disease at screening after second documented CR; OR
      * Flow cytometric confirmation of relapsed T-ALL of at least 0.1% after second CR documented to have been MRD negative < 0.1%; OR
      * Any detectable relapsed disease post-allogeneic HSCT with flow cytometric confirmation of T-ALL of at least 0.1%; OR
      * Biopsy confirmed evidence of relapsed T-LL on lymph node biopsy after second CR; OR
      * Any detectable disease post-allogeneic transplant with biopsy confirmed evidence of T-LL on lymph node biopsy
   2. Refractory disease, defined as:

      * Primary refractory T-ALL or T-LL, defined as failure to achieve CR after induction chemotherapy, per investigator assessment and based on biopsy-confirmed evidence of residual T-ALL or T-LL; OR
      * Relapsed, refractory disease, defined as > 5% BM blasts or biopsy-confirmed evidence of residual TLL after 1 course of re-induction chemotherapy for patients who have relapsed after previously achieving a CR NOTE: Patients with mixed phenotype acute leukemia with T-cell dominant phenotype may be enrolled if the aforementioned criteria are met.
4. Eligible for myeloablative conditioning for and allogeneic HSCT based on the investigator's assessment with an available donor identified by a FACT accredited transplant center.

Key Exclusion Criteria:

1. CNS involvement meeting any of the following criteria: CNS-3 disease, progressive CNS involvement despite therapy, CNS parenchymal or cranial nerve lesions on imaging.
2. Clinically active CNS dysfunction or known history of irreversible neurological toxicity related to prior antileukemic therapy.
3. Receipt of prior CD7 targeted therapy.
4. Systemic antileukemic therapy intended to induce or maintain remission within 14 days prior to completion of screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) and treatment-related adverse events, including serious adverse events (SAEs) and dose-limiting toxicities (DLTs; in Phase 1 only) | Through study completion, an average of 25 months
Overall response rate as defined as proportion of T-ALL patients achieving complete response (CR) or complete response with incomplete hematologic recovery (CRi) or T-LL patients achieving CR or PR at any point after BEAM-201 infusion | From treatment with BEAM-201 through study completion

SECONDARY OUTCOMES:
Proportion of patients who achieve MRD negative response (defined as < 0.1%) by flow cytometry or next generation sequencing (NGS) in patients achieving morphologic response | Starting at Day 28 and multiple time points up to Month 24
Proportion of patients treated with BEAM-201 deemed appropriate for HSCT based on investigator assessment of clinical response | Through study completion, an average of 25 months
Duration of Response (DOR) | Through study completion, an average of 25 months
Relapse-free survival (RFS) | Through study completion, an average of 25 months
Overall survival | Through study completion, an average of 25 months
Relapse-related mortality | Through study completion, an average of 25 months

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Stanford University School of Medicine, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - The University of Kansas Cancer Center, Fairway, Kansas
  - Dana Farber and Boston Children's Hospital, Boston, Massachusetts
  - Cleveland Clinic- Taussig Cancer Center, Cleveland, Ohio
  - OHSU Knight Cancer Institute Hematology Oncology, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Sarah Cannon- TriStar Bone Marrow Transplant, Nashville, Tennessee
  - Methodist Hospital - Texas Transplant Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No